CLINICAL TRIAL: NCT03241134
Title: Changes in Surface Electromyographic Activity of the Upper Trapezius After Dry Needling, Compared to Sham Needling, in Office Workers With Work-related Trapezius Myalgia.
Brief Title: Changes in Surface EMG Activity After Dry Needling Compared to Sham Needling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 01N04215
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Neck Pain, Posterior; Work-Related Condition
Keywords: Dry needling; Sham needling; Office workers; Myofascial pain; Surface electromyography
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): A single dry needling session will be performed with the subject lying on the non painful side. After palpation of a taut band, and detection of a MTrP in the upper trapezius muscle, a trained physiotherapist will penetrate the needle into skin surface, fascia, into the muscle tissue at the MTrP location, and will move the needle up and down in multiple directions. In case local twitch responses are elicited, this will be repeated until the local twitch responses are extinct.
  Interventions: Other: Dry needling
- Sham needling (Sham Comparator): A single sham needling session will be performed with the subject lying on the non painful side. After palpation of a taut band, and detection of a MTrP in the upper trapezius muscle, a trained physiotherapist will penetrate the needle into the skin surface at the MTrP location. The fascia and muscle tissue will not be penetrated.
  Interventions: Other: Sham needling

INTERVENTIONS:
Other: Dry needling — Dry needling (DN) is a myofascial treatment technique, in which a thin, solid filiform needle is inserted directly into the MTrP. During dry needling, local twitch responses (LTR) can be elicited. These are involuntary contractions of muscle fibers, leading to muscle relaxation, an increase in blood flow,recovery of the muscle metabolism and thus a reduction of pain and stiffness.
  Arms: Dry needling
Other: Sham needling — During sham needling, a solid, filiform needle is inserted in the skin surface at the trigger point location, without penetrating the fascia and muscle tissue.
  Arms: Sham needling

SUMMARY:
An experimental study will be conducted to evaluate the effect of a single dry needling session, compared to a sham needling session, on surface EMG activity (signal amplitude and frequency) and pain of the upper trapezius muscle, in office workers with trapezius myalgia.

DETAILED DESCRIPTION:
Neck-shoulder pain is a prevalent problem in office workers. These complaints are often related to myofascial dysfunctions of neck and shoulder muscles, in which the upper trapezius is a vulnerable victim due to prolonged static postures, repetitive upper limb movements and stress, often present during office and computer work. Myofascial dysfunction of the upper trapezius muscle is often referred to as "trapezius myalgia (TM)". Trapezius myalgia is clinically diagnosed with the presence of pain, palpable stiffness and tenderness of the upper part of the trapezius muscle. Several studies show that myofascial trigger points (MTrPs) play an important role in the development and maintenance of myofascial pain and trapezius myalgia. Myofascial trigger points are defined as hyperirritable nodules in a contracture of skeletal muscle fibers, which can cause pain symptoms, motor symptoms as well as autonomic symptoms.

The pathophysiology of MTrPs is still unclear but several hypotheses exist. The most plausible explanation is that, due to sustained postures or repetitive low-level tasks, a sustained irritation of motor end plates with an excessive release of acetylcholine arises. This may lead to a persistent sarcomere contraction, leading to an impaired local blood circulation, a reduced tissue oxygenation and energy depletion, the sensitisation of nociceptors and thus the development of pain.

Dry needling (DN) is a myofascial treatment technique, which has been gaining interest in recent years. During dry needling, a thin, solid filiform needle is inserted directly into the MTrP. During this treatment, local twitch responses can be elicited. These are involuntary contractions of muscle fibers, leading to muscle relaxation, an increased local blood flow, recovery of the muscle metabolism and thus a reduction of pain and stiffness.

In this experimental study, 60 office workers with trapezius myalgia are recruited from several work places with predominantly computer based tasks. Participants are required to perform at least 20 hours of computer work a week, and this since at least one year. Participants are included based on online questionnaires, a clinical examination of neck and shoulder, and the identification of a MTrP in the upper trapezius muscle. All participants will receive information and have to sign an informed consent form.

Participants will be subjected to baseline assessment, which involves measurements of the surface EMG activity (during rest ) and pain scores. Then, subjects will be required to perform a computer task during 20 minutes, surface EMG activity will be measured every 5 minutes. After this computer task, surface EMG activity (during rest ) and pain scores will be measured again. Then, participants will be randomly allocated to either a dry needling group or a sham needling group. The dry needling group will receive a dry needling treatment at the identified trigger point location of the upper trapezius, whereas the sham needling group will receive an intervention in which the needle only penetrates the skin but not the fascia and muscle tissue. After the treatment, surface EMG activity and pain scores will be measured again immediately after, 15 minutes and 30 minutes after completion of the intervention. Thereafter, pain scores will be asked daily, during 7 days after completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Performing office work since at least one year
* Performing computer based tasks for at least 20 hours a week
* NRS > or equal to 3/10
* Clinical diagnosis of trapezius myalgia
* Trapezius myalgia is work-related and thus aggravates during working day/ week
* Presence of a trigger point in the upper trapezius muscle

Exclusion Criteria:

* Being in treatment during the study
* Traumatic injuries/surgery to neck and upper limb region
* Signs of cervical nerve root impingement
* Whiplash injury
* Cardiovascular, neurological, life threatening, systemic and metabolic diseases
* Diagnosis of fibromyalgia/chronic fatigue syndrome
* Shoulder pathology
* Coagulation disorders
* Pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
Changes in resting surface EMG activity (amplitude, RMS) of the upper trapezius after dry needling or sham needling as assessed by the EMG Noraxon 16k Telemyo Device: EMG Noraxon 16k Telemyo | Immediately after a typing task of 20 minutes, immediately after dry or sham needling, 15 minutes and 30 minutes after dry or sham needling
  Changes in resting EMG activity (amplitude, Root Mean Square) of the upper trapezius immediately after, 15 minutes and 30 minutes after dry needling, compared to EMG activity after a typing task, will be measured using surface electrodes placed bilaterally at the MTrP location of the upper trapezius. The change in resting surface EMG activity after dry needling will be compared with the change in surface EMG activity after sham needling.
  Resting surface EMG activity will be expressed as a percentage of a submaximal reference contractions of the upper trapezius (% reference contractions)

SECONDARY OUTCOMES:
Changes in surface EMG activity (amplitude, Root Mean Square) of the upper trapezius during a fatiguing typing task of 20 minutes as assessed by the EMG Noraxon 16k Telemyo Device: EMG Noraxon 16k Telemyo | During the typing task, every five minutes EMG activity will be measured for 30 seconds
  Changes in EMG activity (amplitude, Root Mean Square) of the upper trapezius during a typing task of 20 minutes, will be measured by using surface electrodes placed bilaterally at the MTrP location of the upper trapezius.
  EMG activity during this typing task will be expressed as a percentage of submaximal reference contractions of the upper trapezius (% reference contractions).
Changes in pain score after dry needling, compared to sham needling, as assessed by the numeric rating scale | Immediately after a typing task of 20 minutes, immediately after dry or sham needling, 15 minutes after dry or sham needling, 30 minutes after dry or sham needling, daily during the seven days following the treatment
  Subjects will have to report their actual pain complaints on a numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst pain) after a typing task, immediately after dry or sham needling, 15 minutes after dry or sham needling and 30 minutes after dry or sham needling. In the 7 days following the treatment, pain scores will be asked daily to the participants.
Changes in pain score after a typing task of 20 minutes as assessed by the numeric rating scale | Immediately before and after a typing task of 20 minutes
  Subjects will have to report their actual pain complaints on a numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst pain) before and after a typing task of 20 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Cagnie, PhD, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Meulemeester K, Calders P, Cagnie B. Exploring the Underlying Mechanisms of Action of Dry Needling: What Is the Immediate Effect on Muscle Electrophysiology? An Experimental Randomized Controlled Trial. Am J Phys Med Rehabil. 2022 Jan 1;101(1):18-25. doi: 10.1097/PHM.0000000000001732. PMID 34915542